CLINICAL TRIAL: NCT03570307
Title: Fertility and Obstetric Outcomes After Medical Management Versus Surgical Treatment for First-trimester Miscarriage
Brief Title: Fertility and Obstetric Outcomes After Medical Management Versus Surgical Treatment for First-trimester Miscarriage First-trimester Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, director r&d, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0360-17
Record Dates: First submitted 2018-06-17; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Medical; Abortion, Fetus
Keywords: MISCARRAGE, CURATTAGE MISOPROSTOL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug treatment (Other): Misoprostol for uterine evacuation
  Interventions: Other: medical VS surgical evacuation of the uterus
- surgical treatment (Other): dilatation and curettage for uterine evacuation
  Interventions: Other: medical VS surgical evacuation of the uterus

INTERVENTIONS:
Other: medical VS surgical evacuation of the uterus — mentioned above

SUMMARY:
Study Objective: To compare the time to new pregnancy and pregnancy outcomes in women who received Misoprostol for uterus evacuation versus those treated surgically with dilatation and curettage.

Study Population: Women to be admitted to the Lis maternity department for first trimester failed pregnancy. Patients will choose between medical versus surgical management. Of this group, women interested and successful in achieving a new pregnancy without first engaging in birth control methods will be included in our study.

Inclusion Criteria: Women with first trimester failed pregnancy (up until week 12 according to LMP and up to CRL compatible with 11 gestational weeks) Exclusion Criteria: Women under the age of 18 or over the age of 45, women who conceived via fertility treatments, women with a molar pregnancy.

Study Type: prospective study. Study Description: Women who visit the emergency department or gynecology clinic with a first-trimester miscarriage will be questioned regarding their subsequent family planning. In the event that the woman is interested in another pregnancy, and is not planning to use birth control methods prior to conception, the use of folic acid will be recommended, and she will receive an explanation of the research process. Women who agree to participate in the study orally and who sign a written consent form will be included in the study.

Three to six months following uterine evacuation, study participants will receive a telephone call to assess whether they have conceived, and the case that they had not yet conceived, will receive a follow-up call after an additional three to six months.

Each woman who conceived, will receive a follow-up call to assess the details of the birth. In the event that she did not give birth in the Lis Maternity Hospital, she will be asked to fax a copy of the release letter she received from the hospital.

Type of Birth: Normal vaginal delivery, operative delivery, cesarean section. Birth details will be collected via the automated system in Lis in the event that the birth took These women will be included in the study and will be divided into two groups: surgical vs. medical management. The study will include roughly 200 women in each of the two groups.

It will be clarified that:

1. The researcher will confirm the identity of the participant at the outset of the telephone call.
2. The researcher will request consent and introduce him or herself as a member of the research team from the Lis Hospital. In the event of refusal to participant, the research will apologize and terminate the telephone call.

Study Parameters: 1 .Demographic Parameters of the two groups - age, gravity, parity, ethnicity, history of infertility.

2. Comparison of the success of the surgical treatment versus medical management - in this case, failure is defined as the need for subsequent surgical treatment. This will include data on the percentage of women who received multiple doses of Misoprostol.

3. A comparison of the time (in months) until a new pregnancy is conceived (from the data of the dilatation and curettage or the first dose of the Misoprostol) 4. Pregnancy Outcomes - first trimester miscarriage, obstetric outcomes, early deliveries, pregnancy complications - IUGR, placental abruption, pre-eclampsia, cesarean sections, neonatal outcomes. This data will be collected in multiple telephone conversations - three months after conception and following the delivery date.

1. Validation of details of pregnancies that ended in miscarriage - was the pregnancy desired? Mode of conception (if fertility treatments - which?), months until conception, gestational age at the time that a non-viable pregnancy was diagnosed, mode of pregnancy termination. The details will be validated in relation to details in our automated system.
2. At what month did the woman resume menstruation? Was an ultrasound performed to assess uterine evacuation prior to a new pregnancy conception?
3. Details on pregnancy following dilatation and curettage - time to conception from pregnancy termination, pregnancy outcomes, gestational age at birth (or miscarriage), birth weight, Apgar scores, pH (if available).
4. Data on fertility, age, obstetric history, time to conception of new pregnancies, need for fertility treatments.

Mechanism of Anonymity:

The primary researcher will be responsible for the removal of identifying data. After this data has been removed, in the event that it is still necessary to complete data on the participants, we will make contact with the participant and he will sign a telephone consent form regarding this data completion. In the event that no data is mission and/or after the data is completed through a telephone call, the identifying details will be removed in a way that it will be impossible to replace them. And the telephone consent forms will be saved in a cabinet that can be accessed only by the primary and secondary researchers.

ELIGIBILITY:
Inclusion Criteria:

* Criteria: Women with first trimester failed pregnancy

Exclusion Criteria:

* Women under the age of 18 or over the age of 45, women who conceived via fertility treatments, women with a molar pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Time from evacuation of the uterus to new conception | 2 years

SECONDARY OUTCOMES:
pregnancy outcome | 2 years
  abortion/preterm labor/ term labor